CLINICAL TRIAL: NCT05428735
Title: An International Multicenter Randomized Controlled Trial to Compare Combined Portal and Hepatic Vein Embolization (PVE/HVE) with PVE Alone in Patients with Colorectal Liver Cancer Metastases (CRLM) and a Small Future Liver Remnant (FLR)
Brief Title: The DRAGON 2 Trial
Acronym: DRAGON 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL80303.068.22
Record Dates: First submitted 2022-02-01; First posted 2022-06-23 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer Liver Metastases (CRLM); Small Future Liver Remnant (FLR)
MeSH Terms: interventions — Embolization, Therapeutic

STUDY DESIGN:
Intervention Model Description: 1:1 Randomization between control and interventional group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Portal Vein Embolization (PVE) alone - (control arm) (Active Comparator): Portal Vein Embolization (PVE) alone
  Interventions: Procedure: Embolization
- Combined Portal and Hepatic Vein Embolization (PVE/HVE) - (interventional arm) (Experimental): Combined Portal and Hepatic Vein Embolization (PVE/HVE) - (interventional arm)
  Interventions: Procedure: Embolization

INTERVENTIONS:
Procedure: Embolization — Portal Vein embolization with Glue by a transhepatic approach vs. PVE and Hepatic Vein Occlusion with Vascular plugs via a transjugular or transfemoral approach in the same session as the PVE procedure

SUMMARY:
In the randomized controlled DRAGON 2 trial study subjects will be randomized between two arms, PVE alone (control group) and PVE/HVE (interventional group).

DETAILED DESCRIPTION:
Resection of liver metastases from colorectal cancer (CRLM) improves survival compared to chemotherapy alone and may lead to cure in up to 40% of patients. Extended liver resections are sometimes necessary to resect primarily unresectable/ potentially resectable (PU/PR) colorectal liver metastases. These resections are generally performed if the volume of the future liver remnant (FLR) comprises at least 30% of the total volume of the liver (without the volume of the metastases) or when liver function of the FLR on technetium-99m (99mTc) scintigraphy exceeds 2.67%/min/m2.

When this liver volume or function criterion is not met, a high chance of post-hepatectomy liver failure exists. To prevent this, the induction of liver regeneration between a two-stage hepatectomy is commonly performed.

The current standard procedure to induce regeneration is the embolization of the portal vein branches to the tumor carrying liver (PVE) to induce hypertrophy of the remaining part of the liver which will serve as the FLR. Recently, combined embolization of both portal and hepatic veins (PVE/HVE) has been described as a possible superior alternative to PVE, as it increases and accelerates hypertrophy of the FLR. PVE/HVE combines simultaneous embolization of the main portal vein branches into the tumor carrying liver and the hepatic vein draining this part of the liver. Preclinical studies in pigs, several retrospective studies, and the prospective DRAGON 1 interim analysis (n=60) have demonstrated the safety and feasibility of this novel technique. However, no international randomized controlled trial has been performed, in which combined PVE/HVE is compared with PVE

ELIGIBILITY:
Inclusion Criteria:

* Patients with primarily unresectable/ potentially resectable CRLM with a FLR <30% (<40% in chemotherapy damaged livers)
* Patients with non-resected primary CRC may be included if there is an intention to resect the CRC after the liver treatment (liver first approach) or simultaneously during one of the liver procedures.
* Patients with resectable or ablatable lung or brain metastases can be included (statement about the resectability of these extrahepatic metastases by a tumor board needs to be available)
* 18 Years and older
* Men and women
* Able to understand the trial and provide informed consent.

Exclusion Criteria:

* Pregnant or lactating female.
* Premenopausal females not able or willing to commit to oral contraception
* Patients with prohibitive comorbidities, decision made by local team
* Any patient with non-resectable or non-ablatable extrahepatic disease
* Patients with hepatic malignancies other than CRLM
* Progression of disease by RECIST criteria after cytoreduction chemotherapy
* Complete response after conversion chemotherapy
* Staging CT and (if indicated) CT/MRI brain that demonstrates non-resectable extrahepatic disease
* The anatomy of the liver or manifestation of tumors in relation to the liver veins prohibits the use of combined PVE/HVE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Volume sufficient for resection at week 3 after the embolization | 3 weeks
  Volume sufficient for resection will be based on the first week or third week CT/MR Volumetry. Vauthey calculation for TLV will be used and the FLR volume will be measured centrally (objective panel)
5-year Overall Survival | 5 years
  survival data will be recorded up to 5-years.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M. van Dam, PhD, Principal Investigator — Maastricht Universitair Medisch Centrum
Locations (24):
- Yale New Haven Hospital, New Haven, Connecticut, United States
- Monash Medical Centre, Clayton, Victoria, Australia
- Social Medical Center, South, Vienna, Vienna, Austria
- Belgium (4):
  - Hôpital Erasme, Brussels, Brussels Capital
  - CHU de Liège, Liège, Liège
  - CHU-UCL Namur site Godinne, Yvoir, Namen
  - UZ Gent, Ghent, Oost-Vlaanderen
- Canada (5):
  - Vancouver Coastal Health, Vancouver, British Columbia
  - Juravinski Hospital and Cancer Centre, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - McGill University Health Center, Montreal
- IRCCS San Raffaele Hospital, Milan, Italy
- Netherlands (7):
  - Maastricht University Medical Center+, Maastricht, Limburg
  - Amsterdam UMC, location AMC, Amsterdam, North Holland
  - University Medical Center Groningen, Groningen, Provincie Groningen
  - Erasmus Medical Center, Rotterdam, South Holland
  - Amphia, Breda
  - Maxima Medisch Centrum, Eindhoven
  - Universitair Medisch Centrum Utrecht, Utrecht
- Sweden (2):
  - Linköping University Hospital, Linköping
  - Karolinska University Hospital, Stockholm
- Switzerland (2):
  - Claraspital & Clarunis University Hospital Basel, Basel, Canton of Basel-City
  - Kantonsspital Winterthur (KSW), Winterthur

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication
Access Criteria: Proposal accepted by the DRAGON Collaborative Scientific Committee